CLINICAL TRIAL: NCT05025202
Title: Blood Pressure and Cardiac Autonomic Adaptations to Isometric Exercise Training: a Randomised Sham-controlled Study
Brief Title: Blood Pressure and Cardiac Autonomic Adaptations to Isometric Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18/SAS/47C
Record Dates: First submitted 2021-08-16; First posted 2021-08-27 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants in the sham intervention group were not aware they they were not performing the IET intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IET (Experimental): Participants allocated to this arm performed 4 weeks of isometric wall squat exercise training, 3 times per week.
  Interventions: Other: Isometric exercise training
- Sham (Sham Comparator): Participants allocated to this arm performed 4 weeks of isometric wall squat training, but the training prescription was intentionally provided at an insufficient intensity to achieve any physiology stimulus.
  Interventions: Other: Isometric exercise training
- No intervention control (No Intervention): Participants allocated to this arm did not perform any exercise and were required to maintain usual daily habits.

INTERVENTIONS:
Other: Isometric exercise training — A form of exercise involving static contraction against a wall, sustained for 2 minutes x4 sets per session. 3 sessions a week were required. The intensity was designed to achieve 95% of the participants maximum heart rate.
  Arms: IET; Sham

SUMMARY:
A randomized, sham-controlled intervention measuring the effects of isometric exercise training (IET) on blood pressure and cardiac autonomics.

IET has been proven effective in a plethora of randomized trials, but very little research has employed a sham-controlled design. This researched involved the recruitment of 30 participants who completed a 4 week IET intervention, sham control of the IET intervention, or a non-intervention control period. Pre and post blood pressure and cardiac autonomic measures were acquired and analysed.

The hypothesis of this trial was a significant effect of IET on blood pressure, with no such effects following the sham control or normal control interventions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy with no significant health conditions contraindicating exercise
* Over 18 years of age
* Physically inactive

Exclusion Criteria:

* Achieving current physical activity guidelines
* Abnormal resting ECG
* under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
Blood pressure (systolic, diastolic and mean BP) | At the start of the intervention (pre 4 week intervention)
  Resting office blood pressure measured at brachial artery
Blood pressure (systolic, diastolic and mean BP) | At the end of the intervention (post 4 weeks)
  Resting office blood pressure measured at brachial artery
Cardiac autonomics measured at HRV | At the start of the intervention (pre 4 week intervention)
  LF and HF power spectral measures
Cardiac autonomics measured at HRV | At the end of the intervention (post 4 weeks)
  LF and HF power spectral measures

SECONDARY OUTCOMES:
continuous 5-minute blood pressure (systolic, diastolic and mean BP) | At the start of the intervention (pre 4 week intervention)
  5 minute mean of resting blood pressure measured beat-to-beat
continuous 5-minute blood pressure (systolic, diastolic and mean BP) | At the end of the intervention (post 4 weeks)
  5 minute mean of resting blood pressure measured beat-to-beat

CONTACTS AND LOCATIONS:
Locations (1):
- Canterbury Christ Church University, Canterbury, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Decaux A, Edwards JJ, Swift HT, Hurst P, Hopkins J, Wiles JD, O'Driscoll JM. Blood pressure and cardiac autonomic adaptations to isometric exercise training: A randomized sham-controlled study. Physiol Rep. 2022 Jan;10(2):e15112. doi: 10.14814/phy2.15112. PMID 35083878